CLINICAL TRIAL: NCT07402941
Title: Evaluation of Cochlear (Promontory) Stimulation During Awake Ear Surgery (TONES Study)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Auricle Health Inc. (Industry)
Collaborators: The Cleveland Clinic (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: CLN-0001
Record Dates: First submitted 2025-08-12; First posted 2026-02-11 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Hearing Disorder
Keywords: Hearing; Cochlea
MeSH Terms: conditions — Hearing Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- Electrical extracochlear stimulation (Experimental): Electrical extracochlear stimulation and psychoacoustic testing
  Interventions: Device: Electrical extracochlear stimulation

INTERVENTIONS:
Device: Electrical extracochlear stimulation — Delivery of electrical extracochlear stimulation using electrodes on the middle ear surface. Real-time feedback from subjects on tolerability and auditory percepts

SUMMARY:
The goal of this clinical trial is to learn if short electrical signals can be heard in adult subjects who are otherwise having surgery on their ear.

The main question it aims to answer is:

Can an individual accurately hear different frequencies resulting from the short electrical signals?

DETAILED DESCRIPTION:
The goal of this interventional clinical study is to investigate the feasibility for minimally invasive electrical stimulation of the cochlea as a mechanism for hearing restoration. The main aims of the study are to:

Establish comfortable and tolerable auditory thresholds Investigate the relationship between the position of stimulation, the stimulation parameters and the perceived frequency of any auditory sensation.

This study will enroll patients undergoing middle ear surgery where a brief study procedure will be performed during the course or their surgery. Participants will provide real-time feedback on any auditory sensations and percepts.

ELIGIBILITY:
Inclusion Criteria:

1. Individual is ≥ 18 years old at the time of consent.
2. Individual is scheduled for awake ear surgery that will expose the middle ear (subannular tympanostomy tube placement, tympanoplasty, stapes surgery).
3. Individual is willing to complete intraoperative assessments of promontory stimulation.

Exclusion Criteria:

1. Individual has had severe-to-profound hearing loss for more than 30 years.
2. Individual has congenital hearing loss (for the purpose of this study, onset prior to 2 years of age)
3. Ear canal will not accommodate a speculum with minimum outer diameter (OD) of 4.0 mm or other anatomic challenges present as determined by the study investigator
4. Hearing loss or auditory processing disorder of neural or central origin
5. Active middle ear infection
6. History of cholesteatoma treated within the past 2 years
7. Ossification of the cochlear or other previously identified cochlear anomaly
8. Prior major head trauma (stroke, hemorrhage, traumatic brain injury) within past 2 years
9. Contralateral presence of cochlear implant
10. Individual is pregnant.
11. Individual is unable or unwilling to complete training for qualitative evaluation of promontory electrical stimulation.
12. A disability that could interfere with intraoperative evaluations as determined by study investigator.
13. Profound tinnitus
14. History of vertigo that would interfere with the planned investigation as determined by the principal investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2025-06-02 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Stimulation discrimination | Time of study procedure
  Accuracy of comparison of paired stimulation presentations as indicated by subject. This will be measured using a same-different task, where two stimulation paradigms are compared. The participant will be presented two consecutive stimuli, randomized to be the same or different. The participant will verbalize whether they felt the stimuli were the same or different. This will be repeated five times and graded on a percentage scale.

SECONDARY OUTCOMES:
Threshold and most comfortable level | Time of study procedure
  Stimuli will be presented at different positions on the cochlear promontory. For each position the current applied will be gradually increased in small increments from zero. The current threshold at which the stimulus is first detected by the participant will be recorded. The current level will then be increased to a level at which the participant reliably and comfortably detects the stimulus which will be recorded as the Most Comfortable Level (MCL).
Stimulation effects | Time of study procedure
  The subject will ask the participant to report any new sensations or discomfort experienced during the stimulation. The investigator will also be monitoring the patient for signs of discomfort or off-target nerve stimulation such as facial twitching. These effects will be recorded with the stimulation parameters and location used.

CONTACTS AND LOCATIONS:
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No